CLINICAL TRIAL: NCT03581162
Title: Atherosclerosis in Juvenile Mixed Connective Tissue Disease
Brief Title: Atherosclerosis in Juvenile Mixed Connective Tissue Disease (ACTID)
Acronym: ACTID
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Karolina Ryeng Skagen, Doctor/PostDoc, Oslo University Hospital
Other Study IDs: 2012/1721
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Ultrasonography, Carotid Arteries; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with diagnosis of Juvenile Mixed Connective Tissue Disease
  Interventions: Diagnostic Test: Carotid Ultrasound and venous blood sampling
- Controls: Healthy, age-and sex-matched controls
  Interventions: Diagnostic Test: Carotid Ultrasound and venous blood sampling

INTERVENTIONS:
Diagnostic Test: Carotid Ultrasound and venous blood sampling — Carotid ultrasound and blood sampling

SUMMARY:
This Study investigates presence of preclinical atherosclerosis in patients with Juvenile Mixed Connective Tissue Disease in Norway.

DETAILED DESCRIPTION:
Patients and controls are examined with carotid ultrasound, venous blood is drawn, and they undergo a clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MIxed Connective Tissue Disease

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosis of Juvenile Mixed Connective TIssue Disease in Norway
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Presence of carotid atherosclerosis | 20 minutes
  measuring intima-media thickness

SECONDARY OUTCOMES:
blood markers of endothelial dysfunction | 20 minutes

IPD SHARING:
Plan to Share IPD: No